CLINICAL TRIAL: NCT06590493
Title: Doxecitine and Doxribtimine-Expanded Access
Status: Available | Type: Expanded Access
Sponsor: UCB BIOSCIENCES, Inc. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Other Study IDs: doxecitine and doxribtimine-EA
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Thymine Kinase 2 Deficiency
Keywords: Thymine Kinase 2 Deficiency; TK2; TK2d

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: doxecitine and doxribtimine — TK0113 and TK0115: Doxecitine and doxribtimine is dosed daily and will be administered orally or via feeding tube. The patient may continue to receive doxecitine and doxribtimine treatment within the EAP as long as the benefit / risk balance remains positive in the opinion of the treating physician or access to commercially available doxecitine and doxribtimine, when it becomes available.

SUMMARY:
This Expanded Access Record for doxecitine and doxribtimine includes the following managed access programs and status:

TK0113: Available TK0115: Available

DETAILED DESCRIPTION:
TK0113: Data Collection for Patients in the Company Supported Expanded Access Program TK0115: TREATMENT PROTOCOL FOR DOXECITINE AND DOXRIBTIMINE - Company-sponsored Intermediate-size Cohort Expanded Access Program for Doxecitine and Doxribtimine for Patients with Thymidine Kinase 2 Deficiency (TK2d) with an Age of Symptom Onset ≤ 12 Years

ELIGIBILITY:
Inclusion Criteria:

TK0113:

* Pediatric and adult patients with a diagnosis of TK2d based on confirmed reportable variant(s) in the TK2 gene in countries where UCB has an affiliate/local safety officer Signs and symptoms compatible with TK2d disease
* Risk of major disability or death resulting from TK2d
* The patient must be willing to receive treatment with doxecitine and doxribtimine via this program, which includes signing an authorization form for sharing genetic test results, medical data and other related information with UCB, its third-party agents and health authorities
* The patient/legal guardian or representative has given informed consent (and age-appropriate assent) to treatment prior to administering doxecitine and doxribtimine in a manner consistent with all national requirements. This also includes consent for the transmission of a copy of the anonymized data, such as serious adverse event (SAE) and pregnancy reports (in compliance with local regulatory authority requirements) to UCB third-party agents where allowable by local regulations and to the country regulatory authority as required.
* The patient does not qualify for or is unable to participate in a UCB sponsored ongoing clinical trial evaluating doxecitine and doxribtimine.

TK0115:

* Diagnosis of TK2d based on confirmed reportable variant(s) in the TK2 gene
* Age of TK2d symptom onset ≤ 12 years
* The patient or care provider must be willing to receive treatment with doxecitine and doxribtimine via this program
* Patient has consented to the contraception, pregnancy, and lactation requirements where relevant
* The patient does not qualify for or is unable to participate in a UCB-sponsored clinical trial evaluating doxecitine and doxribtimine for the treatment of patients with TK2d

Exclusion Criteria:

TK0113:

* Confirmed diagnosis of other genetic or polygenic disease likely to confound clinical presentation of TK2 deficiency
* Patient has a hypersensitivity to any of the excipients in doxecitine and doxribtimine
* Inability to tolerate oral or gastric tube administration of doxecitine and doxribtimine
* History of liver disease, or liver function test results (alanine aminotransferase[ALT], aspartate transaminase [AST], or total bilirubin) ≥3× upper limit of normal at Screening without prior Sponsor approval
* Patients with elevated transaminases (ALT, AST > 3xupper limit of normal) without increase in bilirubin should be further evaluated to exclude other causes of liver injury and may be enrolled with UCB approval or may be rescreened
* Renal insufficiency requiring dialysis
* Discontinuation of prior nucleos(t)ide treatment for TK2d because of adverse event(s)
* Any other concurrent inborn errors of metabolism
* Severe end-organ hypo-perfusion syndrome secondary to cardiac failure resulting in lactic acidosis
* Patient has a medical or any other extenuating condition or circumstance that may, in the opinion of the investigator, pose an undue safety risk to the patient or compromise his/her ability to comply with, or adversely impact, protocol requirements
* Concurrent participation in another interventional trial or named patient program where investigational drug is received
* Any other reason that UCB may determine that the patient is unsuitable for named patient / compassionate use of doxecitine and doxribtimine

TK0115:

* History of liver disease or liver function test results (alanine aminotransferase [ALT], aspartate transaminase [AST], or total bilirubin) ≥ 3 × upper limit of normal (ULN) at Baseline or bilirubin > 1.5 × ULN. Isolated bilirubin > 1.5 × ULN is acceptable if bilirubin is fractionated and direct bilirubin < 35%
* Patients with elevated transaminases (ALT and/or AST > 3 × ULN) without increase in bilirubin should be further evaluated to exclude other causes of liver injury and may be enroled with UCB approval
* Patient has a medical, mental, or any other extenuating condition or circumstance that may, in the opinion of the treating physician, pose an undue safety risk to the patient or compromise his/her ability to comply with, or adversely impact, protocol requirements
* Renal insufficiency requiring dialysis
* Discontinuation of prior nucleoside treatment for TK2d due to adverse event(s) (AEs)
* Concurrent participation in another interventional trial or named patient program where investigational drug is received
* Known hypersensitivity to doxecitine and doxribtimine or any excipients of the drug substance (silicon dioxide and magnesium stearate)
* Inability to tolerate oral or enteral feeding tube administration of doxecitine and doxribtimine
* Female patients will not be eligible to participate if they are pregnant, plan to become pregnant during the course of the program, or are breastfeeding

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273